CLINICAL TRIAL: NCT01228552
Title: A Randomized Double Blind, Placebo Controlled Phase III Trial to Determine the Efficacy and Safety of Topical Intra-oral Ketoprofen for the Treatment of Acute Migraine
Brief Title: The Efficacy and Safety of Intra-oral Topical Ketoprofen for the Treatment of Acute Migraine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Behar, Caren, M.D. (Individual)
Responsible Party: Behar, Caren M.D., New York Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 79,629
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-10

CONDITIONS: Migraine Disorders; Migraine Headache; Migraine; Acute Migraine
Keywords: Acute Migraine Treatment; Migraine Treatment; Migraine; Headache; Treatment
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical, intra-oral ketoprofen gel (Active Comparator)
  Interventions: Drug: Topical, intra-oral ketoprofen gel
- Placebo gel (Placebo Comparator)
  Interventions: Other: Placebo gel

INTERVENTIONS:
Drug: Topical, intra-oral ketoprofen gel — Ketoprofen gel will be applied, using a cotton applicator, to the gingival mucosa at the onset of migraine. A second application may be used at 20 minutes, if necessary.
  Arms: Topical, intra-oral ketoprofen gel
Other: Placebo gel — Placebo gel will be applied, using a cotton applicator, to the gingival mucosa at the onset of migraine. A second application may be used at 20 minutes, if necessary.
  Arms: Placebo gel

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intra-oral topical ketoprofen for the treatment of acute migraine.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Migraine as per IHS with aura
* Established diagnosis of Migraine as per IHS without aura
* At least 2 migraines per month
* At least 18 years of age

Exclusion Criteria:

* Pregnancy or Lactation
* Other Headache Conditions including basilar, hemiplegic, or ophthalmoplegic migraines
* Chronic Daily Headache
* Allergy or Sensitivity to NSAIDs
* Other Severe Medical Conditions including GI bleeding, blood dyscrasias, thrombocytopenia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Pain relief (defined as at least 2 graded reduction in a 5-grade scale) at 120 minutes post-treatment | Within 240 minutes post-treatment

SECONDARY OUTCOMES:
Pain free status at 30, 60, 120, and 240 minutes post-treatment based on headache severities reported in patient's journals | Within 240 minutes post-treatment
Pain relief at 30, 60, and 240 minutes post-treatment based on headache severities reported in patient's journals | Within 240 minutes post-treatment
Relief of Photophobia at 30, 60, 120, and 240 minutes post-treatment | Within 240 minutes post-treatment
Relief of Phonophobia at 30, 60, 120, and 240 minutes post-treatment | Within 240 minutes post-treatment
Relief of Nausea at 30, 60, 120 and 240 minutes post-treatment | Within 240 minutes post-treatment
Relief of Vomiting 30, 60, 120 and 240 minutes post-treatment | Within 240 minutes post-treatment
Need for Rescue Medication between the time of dosing to 240 minutes | Within 240 minutes post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Caren Behar, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States